CLINICAL TRIAL: NCT05417789
Title: A Phase III, Multicentre, Randomised, Double-Blind Study to Assess the Safety and Efficacy of Emactuzumab vs. Placebo in Subjects With Tenosynovial Giant Cell Tumour
Brief Title: Study of Emactuzumab for Tenosynovial Giant Cell Tumor (TGCT)
Acronym: TANGENT
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: SynOx Therapeutics Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SNX-301-020
Record Dates: First submitted 2022-06-01; First posted 2022-06-14 (Actual); Last update posted 2026-02-02 (Actual); Status verified 2025-12

CONDITIONS: TGCT
Keywords: TGCT, Tenosynovial Giant Cell Tumour; PVNS, Pigmented Villonodular Synovitis; Synovitis; Emactuzumab; Local TGCT; Diffuse TGCT
MeSH Terms: conditions — Synovitis, Pigmented Villonodular; Synovitis | interventions — emactuzumab

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Group 1 in Part 1/Part 2: Emactuzumab (Experimental): Group 1: Subjects receiving emactuzumab administered intravenously (i.v) on Day(D)1 and repeated once every two weeks (Q2W) for a total of 5 times, followed by an observation period of 3 months leading to a total period of 24 weeks in Part 1 and continued with a follow-up phase in Part 2. Eligible Subjects assigned to active drug in Part 1 have the option to receive open-label retreatment in Part 2.
  Interventions: Drug: Emactuzumab
- Group 2 in Part 1 and Part 2: Placebo (Placebo Comparator): Group 2: Subjects receiving placebo administered intravenously (i.v) on D1 and repeated once every two weeks (Q2W) for 5 times followed by an observation period of 3 months to a total period of 24 weeks in Part 1. In Part 2, Eligible Subjects will have the option to receive open-label emactuzumab, administered by i.v once every 2 weeks (Q2W) for a total of 5 times.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Emactuzumab — Emactuzumab administered once every 2 weeks (q2w)
  Arms: Group 1 in Part 1/Part 2: Emactuzumab
Drug: Placebo — Matching placebo administered once every 2 weeks (q2w)
  Arms: Group 2 in Part 1 and Part 2: Placebo

SUMMARY:
This is a multicenter, Phase 3, randomised, double-blind, placebo-controlled study, which aims to evaluate the efficacy and safety of the investigational drug emactuzumab for the treatment of patients with localized or diffuse TGCT where surgical removal of the tumor is not viewed as an option.

The study consists of two parts. In Part 1, eligible subjects will be assigned in a 2:1 ratio to receive either emactuzumab or matching placebo in a double-blind fashion, that will be administered in total 5 times as an intravenous (i.v.) infusion once every 2 weeks. This will be followed by an observation period of 3 months leading to a total duration of 24 weeks in Part 1. A number of assessments will be carried out during the course of the study, including physical examinations, blood tests, imaging studies, electrocardiograms, and questionnaires. Part 2 is a long-term double-blind follow-up phase of the subjects on emactuzumab or placebo. Subjects assigned to placebo in Part 1 have the option, subject to eligibility, to crossover to receive open-label emactuzumab in Part 2. Subjects assigned to active drug in Part 1 have the option to receive open-label retreatment under certain circumstances.

ELIGIBILITY:
Inclusion Criteria:

* Age >12 years
* Biopsy-confirmed (standard of care diagnosis history) local or diffuse TGCT where surgical resection would be associated with predicted worsening functional limitations through surgical joint damage, and/or subject has an anticipated high risk of early recurrence as determined by a multidisciplinary tumour board or equivalent, or any other morbidity associated with the surgery, and/or surgical treatment is not expected to improve the clinical outcomes of the subject.
* Measurable disease: longest diameter ≥20 mm.
* Adequate organ and bone marrow function
* If a woman of childbearing potential (WOCBP), must have a negative pregnancy test prior to starting treatment and agree to use a highly effective method of contraception
* Participants must have given written consent

Exclusion Criteria:

* If a female, the subject is pregnant or breast feeding.
* Medical conditions, including auto-immune, requiring systemic immunosuppression. Any systemic treatment for these conditions (eg, glucocorticoids) is not allowed within 4 weeks of Screening and during the study.
* Known metastatic TGCT or other active cancer that requires concurrent or planned treatment
* Received systemic therapy for TGCT (investigational or approved) targeting CSF-1 or CSF-1R or any multi-tyrosine kinase inhibitor (eg nilotinib and imatinib) within 3 months prior to screening
* Any surgery, chemotherapy or radiotherapy within 3 months of screening
* Unresolved clinically significant toxicity from a previous treatment or any history of serious liver toxicity.
* Current or chronic history of liver disease.
* Inadequate renal and liver function
* Systemic antiretroviral therapy within 3 months of baseline
* Within 6 months of baseline has experienced: clinically significant myocardial infarction, severe/unstable angina pectoris, congestive heart failure New York Heart Association (NYHA) Class III or IV, or pulmonary disease (NYHA Criteria 1994) including severe thromboembolic event; incompletely healed clinically significant wounds, including bone fractures; pathological fracture or significant hypercalcaemia.

Min Age: 12 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 128 (Estimated)
Dates: Start 2024-10-09 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Overall Response Rate (ORR) | Day 0 - Day 180 (6 months)
  Objective Response Rate (ORR = complete response [CR] + partial response [PR]) by 6 months from initiation of therapy according to RECIST v1.1 based on independent, blinded central review

SECONDARY OUTCOMES:
Physical Function | up to 24 months
  Change in Patient-Reported Outcomes Measurement Information System Physical Function (PROMIS-PF) TGCT from baseline to 6 months
Range of Motion (ROM) | up to 24 months
  Mean change from baseline in active ROM of the joint over time
Worst Stiffness | up to 24 months
  Mean change from baseline in the Worst Stiffness Numeric Rating Scale (NRS) score over time
Worst Pain | up to 24 months
  Mean change in Pain Numerical Rating Scale (NRS) from baseline over time
Quality of Life (QoL) | up to 24 months
  Change in EuroQol 5-dimension, 5-level questionnaire (EQ-5D-5L)
Duration of response (DoR) | up to 24 months
  Duration of response (DoR) as measured by RECIST version 1.1
Tumour volume score (TVS) | up to 24 months
  Change in Tumour volume score (TVS)
Surgical Intervention Rate | up to 24 months
  The number of subjects who undergo surgery during the study for TGCT

CONTACTS AND LOCATIONS:
Overall Officials: Jean Y Blay, Prof, MD, Principal Investigator — Comprehensive Cancer Centre of Lyon
Locations (48):
- United States (10):
  - NextGen Oncology, Beverly Hills, California
  - Sarcoma Oncology Research Center, LLC, Los Angeles, California
  - USC Norris Comprehensive Cancer Center, Los Angeles, California
  - University of Kansas Cancer Center (Overland Park) - USOR, Overland Park, Kansas
  - University of Minnesota, Minneapolis, Minnesota
  - Duke Cancer Center, Durham, North Carolina
  - The Ohio State University, Columbus, Ohio
  - OHSU Knight Cancer Institute Hematology Oncology, Portland, Oregon
  - MD Anderson Cancer Center, Houston, Texas
  - MedStar Washington Hospital Center, Georgetown, Washington
- LKH-Universitätsklinikum Graz, Graz, Austria
- Belgium (2):
  - Cliniques Universitaires Saint-Luc, Woluwe-Saint-Lambert, Brussels Capital
  - UZ Gent - Department of Medical Oncology, Ghent
- Canada (3):
  - Arthur J.E. Child Comprehensive Cancer Centre, Calgary, Alberta
  - Princess Margaret Cancer Centre, Toronto, Ontario
  - McGill University Health Centre (MUHC), Montreal, Quebec
- France (8):
  - Centre Antoine Lacassagne, Nice, Alpes-Maritimes
  - Institut Bergonie - PPDS, Bordeaux, Gironde
  - Institut de Cancerologie de Ouest - Saint Herblain, Saint-Herblain, Loire-Atlantique
  - AP-HP - Hôpital Cochin - Port-Royal, site Cochin, Paris, Paris
  - Centre Léon Bérard Centre Régional de Lutte Contre Le Cancer Rhône Alpes, Lyon, Rhône
  - UNICANCER - Centre Oscar Lambret, Lille
  - Institut Curie - Hôpital de Paris, Paris
  - Oncopole Claudius Regaud Oncologie Médicale, Toulouse
- Italy (8):
  - Fondazione Policlinico Universitario Campus Bio-Medico, Rome, Lazio
  - Fondazione del Piemonte per l'Oncologia (IRCCS), Candiolo, Piedmont
  - Azienda Ospedaliera Universitaria Policlinico Paolo Giaccone, Palermo, Sicily
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento di Cisanello, Pisa, Tuscany
  - Nuovo Ospedale di Prato, Prato, Tuscany
  - IRCCS lstituto Ortopedico Rizzoli, Bologna
  - Fondazione IRCCS Istituto Nazionale dei Tumori, Milan
  - Azienda Ospedaliero Universitaria Pisana - Stabilimento di Cisanello, Pisa
- Leids Universitair Medisch Centrum, Leiden, Netherlands
- Seoul National University Hospital, Seoul, South Korea
- Spain (6):
  - Hospital Clinico San Carlos, Madrid, Madrin
  - Hospital Universitario Fundacion Jimenez Diaz, Zaragoza, Zaragoza
  - Hospital de La Santa Creu i Sant Pau, Barcelona
  - Hospital Universitario Virgen del Rocio - PPDS, Seville
  - Hospital Universitari i Politecnic La Fe de Valencia, Valencia
  - Hospital Universitario Miguel Servet, Zaragoza
- Skanes Universitetssjukhus Lund, Lund, Skåne County, Sweden
- Switzerland (2):
  - Universitäts Kinderspital Beider Basel (UKBB), Basel
  - Inselspital - Universitätsspital Bern, Bern
- Taiwan (2):
  - National Taiwan University Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- United Kingdom (3):
  - St James's University Hospital, Leeds
  - University College Hospital, London
  - Churchill Hospital, Cancer Haematology Center, Oxford

IPD SHARING:
Plan to Share IPD: No
Summary (synopsis) of the CSR